CLINICAL TRIAL: NCT06353984
Title: Effects of a Nutritionally Balanced In-between Meal Food Product on Cognitive Function in the Elderly - an Explorative Study
Brief Title: Effects of In-between Meal Products on Cognitive Function in the Elderly
Acronym: Minimeal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Minimeal 1.0
Record Dates: First submitted 2024-02-28; First posted 2024-04-09 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Function
Keywords: cognitive function

STUDY DESIGN:
Intervention Model Description: Three-arm randomized controlled trial that includes a double-blinded, two-armed intervention and a non-blinded control arm without any intervention
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators and participants are partly blinded as the control group receives no placebo product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): Intervention group receives the study product
  Interventions: Dietary Supplement: Minimeal product
- Reference group (Active Comparator): Reference group receives a reference product
  Interventions: Dietary Supplement: Reference product
- Control group (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Minimeal product — Intervention product consisting of bioprocessed oats and chickpeas
  Arms: Intervention group
Dietary Supplement: Reference product — Reference product mimicking available soups and fruit drinks
  Arms: Reference group

SUMMARY:
The overall aim of the present 9-week intervention study is to determine how a healthy drinkable in between meal affects cognitive function and brain activity in healthy adults 70 years and older. Secondary, the study also investigates the impact of the intervention on low grade inflammation, immune function, gut health, body composition, physical function, and well-being as secondary or exploratory outcomes. The study products have the potential to lower chronic low-grade inflammation in the elderly, improve nutrition and thereby contribute to healthy aging including cognitive function, and the study will also give additional insight regarding secondary and exploratory outcomes.

DETAILED DESCRIPTION:
The current study is a nine week three-arm randomized controlled trial that includes a double-blinded, two-armed intervention and a non-blinded comparative arm without any intervention. This study will investigate the effects of a healthy in between meal consisting of processed oats and chickpeas on cognitive function and functional brain activity in healthy older men and women 70 years and older (primary endpoints) and explore the effect of the intervention product on blood markers, body composition, physical activity, physical function, and self-reported well-being in the earlier mentioned population (secondary endpoint). Furthermore, the study will give insight in the preventative value of the intervention product on earlier mentioned age-related conditions as well as adherence to the study product and gives guidance towards further research regarding the effect of food product on age related conditions. Participants will visit the study centre at seven occasions, one time before (pre visit) and six times during the study period to perform one or more tests and/or examinations. The pre visit takes place before the baseline, visit 1 and 2 are at baseline, and visit 3 and 4 are the mid-study-visits in week 3 and 6 of the interventional period. Visit 5 and 6 take place at the last interventional week, ie week 9. Data and sample collection takes place as following:

* visit 0: Eligibility screening and informed consent
* Week 1: visit 1 baseline: Body composition, blood samples, fecal samples, questionnaires and physical activity and function, cognitive function
* Week 1: visit 2 baseline fMRI: Structural MRI, RS-(MRI), N-back task fMRI, word recognition task
* Week 3: visit 3 intermediate visit I: Body composition, blood samples, questionnaires, compliance
* Week 6: visit 4 Intermediate visit I: Body composition, blood samples, questionnaires, compliance
* Week 9: visit 5 study end: same procedure as visit 1
* Week 9. Visit 6 study end: same procedure as visit 2

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-related procedure
* Age 70 years and above
* Normal weight to overweight at the screening defined as BMI range 18.5-31.9
* Willing to abstain from regular consumption of medication known to alter gastrointestinal function or inflammatory status after being included and during the study
* Willingness to pick up study products and eat the products according to the instructions each day

Exclusion Criteria:

* Diagnosis of type 1 and/or type 2 diabetes
* Immobile (defined as the inability to participate in all study-related procedures)
* History of complicated gastrointestinal surgery
* Diagnosed inflammatory bowel disease (IBD)
* Current diagnosis of psychiatric disease/s or syndromes
* Current diagnosis of neurodegenerative disease
* Systemic use of antibiotics and/or steroid medication in the last 4 months prior to inclusion
* Use of probiotics, prebiotics, fermented foods, kombucha, and any other product known to modulate gut microbiota composition in the last 2 months prior to inclusion
* Use of any non-steroidal anti-inflammatory drug (NSAID) more than 3 times a week in the last 2 months prior to inclusion
* Use of statins
* Consumption of any NSAID within 7 days of study start
* Any condition which could interfere with intestinal barrier function (e.g. gluten sensitivity, lactose intolerance, celiac disease, IBS, IBD) as decided by the principal investigators' discretion
* Vegetarian diet
* Allergy to ingredients included in either investigational or reference products
* Regular smoking, use of snuff, nicotine, or e-cigarette use
* Drinking more than 9 standard cups of alcohol per week and/or more than 3 standard cups of alcohol per occasion
* Regular use, for more than three times a week for the last 2 months and/or 7 days prior to inclusion, of medications which according to the principal investigator can have an anti-inflammatory effect or affect in any way the intestinal barrier function or have an impact on the study analysis (such as laxatives, anti-diarrheal, anti-cholinergic, etc.)
* After being included in the study, starting any medication or treatment that could potentially influence the study participation and/or study analysis
* Cerebral bleeding or history of cerebral bleeding
* Claustrophobia
* In operated apparatus (e.g., pacemaker)
* Aneurysm clips or shunts in the head
* Grenade-splinter or metal-splinter in the body (e.g., eyes)
* Metal or electrodes in the body (e.g., temp-catheter, aorta stent, cochlea implant)
* Comprehensive tooth-implants or prosthesis
* Operated in the head or in the heart
* Swallowed a video-capsule
* Left-handed
* Severe vision impairments
* Being highly physically active, competing as a master athlete and/or partaking in physical demanding training more than four times per week, extreme exercising
* Any other reason the investigator feels the subject is not suitable for participation in this aspect of the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Functional brain activity | 9 weeks
  Functional brain activity will be measured by functional magnetic resonance imaging (fMRI)) during the n-back task

SECONDARY OUTCOMES:
Fasting blood glucose/insulin | 9 weeks
  Fasting blood glucose insulin will be taken and the HOMA index (Homeostatic Model Assessment for Insulin Resistance) expressed in mmol/L or mg/dL will be used to assess insulin resistance
Blood fats/lipid status | 9 weeks
  Blood fats/lipid status unit of measurement concentration given mmol/L
Interleukin-6 | 9 weeks
  Concentration of interleukin-6 measured in in blood serum corrected for baseline, unit of measurement concentration given as pg/mL
High-sensitivity C-reactive protein | 9 weeks
  High-sensitivity C-reactive protein (HsCRP) measured in blood corrected for baseline, unit of measurement concentration given as mg/L
Tumor necrosis factor | 9 weeks
  Concentration of Tumor necrosis factor (TNF) in blood serum corrected for baseline, unit of measurement concentration given as pg/mL
Interferon-gamma | 9 weeks
  Concentration of Interferon-gamma (IFN-Gamma) in blood serum corrected for baseline, unit of measurement concentration given as pg/mL
Zonulin | 9 weeks
  Zonulin (haptoglobin 2 precursor) is a protein that increases the permeability of tight junctions between cells of the wall of the digestive tract, measured in faeces.
Intestinal fatty-acid binding protein | 9 weeks
  Intestinal fatty-acid binding protein (I-FABP) measured in faeces
Cognitive function | 9 weeks
  Cognitive function will be assessed by an off-line multi-domain cognitive test battery computer-based, word recognition task
Magnetic resonance imaging (MRI) | 9 weeks
  Resting state connectivity functional MRI (rsfMRI) and brain morphology from structural scans (brain and brain stem) are measured by MRI
The Perceived Stress Scale | 9 weeks
  The Perceived Stress Scale (PSS) questionnaire is used to measure the perception of stress in life and has 10 questions with the following options to answer: 0 = Never 1 = Almost Never 2 = Sometimes 3 = Fairly Often 4 = Very Often
Hospital Anxiety and Depression Scale | 9 weeks
  The validated Hospital Anxiety and Depression Scale (HADS) questionnaire will be used to assesses symptoms of depression and anxiety. The HADS has 7 questions related to depressions and 7 questions related to anxiety. A higher total score indicates more depression or anxiety with the following cut off scores: 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
SF 36 | 9 weeks
  The SF 36 (short form) questionnaire is used to assess general health Status. The SF-36 consists of 36 questions. Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to high quality of life
Western Ontario and McMaster Osteoarthritis Index | 9 weeks
  To evaluate hip and knee osteoarthritis Western Ontario and McMaster Osteoarthritis Index (WOMAC) questionnaire is used. The WOMAC is a self-administered questionnaire consisting of 24 items divided into 3 subscales. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. A sum of the scores for all three subscales gives a total score
Clinical Outcomes in Routine Evaluation | 9 weeks
  The translated and validated Swedish version of the Clinical Outcomes in Routine Evaluation (CORE-GP) is used to evaluate psychological wellbeing. The CORE-GP consists of 34 questions about how they have been feeling over the last week, using a 5-point scale (not at all, only occasionally, sometimes, often, most or all the time. The scale covers four dimensions: subjective well-being, problems/symptoms, life functioning, risk/harm
Gastrointestinal Symptoms Rating Scale | 9 weeks
  To assess gastrointestinal symptoms the Gastrointestinal Symptoms Rating Scale (GSRS) questionnaire is used. The questionnaire consists of 15 questions combined into five symptom clusters: reflux, abdominal pain, indigestion, diarrhoea and constipation. Each questions is rated on a 7-point likert scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms
Pittsburgh Sleep Quality Index | 9 weeks
  To assess sleep quality and sleep disturbances over a one-month time interval the Pittsburgh Sleep Quality Index (PSQI) questionnaire is used. Each questionnaire's 19 self reported items belong to one of seven categories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, daytime dysfunction. The questionnaire consists of a combination of likert-type and open-ended questions. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.
International Physical Activity Questionnaire for the Elderly short form | 9 weeks
  The International Physical Activity Questionnaire for the Elderly (IPAQ-E) short form consists of 4 questions regarding time spend sitting, walking, heavy physical activities or sport or very heavy activities or sport
Historical Physical Activity Questionnaire | 9 weeks
  The Historical Physical Activity Questionnaire HAPAQ assesses physical activity behaviour between the age of 20 to 65 years and consists of questions regarding physical activity, sports and labour performed per year, month and average minutes per week
Food frequency questionnaire | 9 weeks
  The Meal-Q Food frequency questionnaire is used to assess if participants have altered dietary patterns during the intervention. The questionnaire consists of 174 questions about foods, dishes and drinks (including alcoholic drinks) as well as pictures of different portion sizes for cooked dishes, questions about meal order, eating behaviour (with regard to restaurant visits, fast food, salad buffets, salt on food, consumption of diet products) and supplements.
Physical activity | Only at baseline (week 1)
  Habitual physical activity will be assessed by accelerometery activity monitor during a week during waking time. Counts per minute are registered and converted into daily average times spent in sedentary behaviour, light-intensity physical activity, and moderate-to-vigorous intensity physical activity.
Muscle mass | 9 weeks
  Muscle mass is assessed with bioelectrical impedance (BIA)
Fat mass | 9 weeks
  Fat mass is assessed with bioelectrical impedance (BIA)
Body mass index | 9 weeks
  Body mass index (BMI) is calculated as weight (in kg)/ height^2 (in m^2)
Waist circumference | 9 weeks
  Waist circumference is measured to the nearest 0.1 cm with a steel tape at the midpoint between iliac crest and lower costal marginBody mass index (BMI)
Aerobic capacity | 9 weeks
  Aerobic capacity is assessed by a maximal walk test on a graded treadmill (Modified Bruce Protocol) where a further stage and time into the stage indicates a better aerobic fitness
Balance | 9 weeks
  Balance by the single leg stance balance test with eyes open and eyes closed where longer time indicates a better balance
30-sec repeated chair raise | 9 weeks
  Lower body muscle performance is assessed by the 30-sec repeated chair raise where more repetitions indicates a better performance
Maximal leg strength | 9 weeks
  Maximal leg strength is assessed by the leg press exercise where a larger amount in kilograms lifted indicates a higher maximal leg strength
Maximal handgrip strength | 9 weeks
  Maximal handgrip strength by the handgrip test where total amount of kilogram or kilogram per bodyweight indicates a higher total, or relative handgrip strength respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University, Örebro, Sweden